CLINICAL TRIAL: NCT00572156
Title: Recombinant Human Growth Hormone (rhGH) and Recombinant Human Insulin-like Growth Factor-1 rhIGF-1) Combination Therapy in Children With Short Stature Associated With IGF-1 Deficiency: A Six-year, Randomized, Multi-center, Open-label, Parallel-group, Active Treatment Controlled, Dose Selection Trial
Brief Title: rhGH and rhIGF-1 Combination Therapy in Children With Short Stature Associated With IGF-1 Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated due to strategic reasons.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS316; 2019-000843-29 (EudraCT Number)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Insulin-like Growth Factor-1 Deficiency
Keywords: IGF-1 Deficiency; growth; ISS; Constitutional growth delay; Primary IGFD; Primary IGF Deficiency
MeSH Terms: conditions — Insulin-Like Growth Factor I Deficiency; Puberty, Delayed | interventions — Human Growth Hormone; mecasermin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1. rhGH Alone (Active Comparator)
  Interventions: Drug: NutropinAq® (Somatropin [rDNA origin])
- 2. Combination Dose (Experimental)
  Interventions: Drug: Increlex® (Mecasermin [rDNA origin] injection) + NutropinAq® (Somatropin [rDNA origin])
- 3. Combination Dose (Experimental)
  Interventions: Drug: Increlex® (Mecasermin [rDNA origin] injection) + NutropinAq® (Somatropin [rDNA origin])
- 4. Combination Dose (Experimental)
  Interventions: Drug: Increlex® (Mecasermin [rDNA origin] injection) + NutropinAq® (Somatropin [rDNA origin])

INTERVENTIONS:
Drug: NutropinAq® (Somatropin [rDNA origin]) — rhGH (Somatropin) 45µg/kg once daily injection
  Other Names: GH
  Arms: 1. rhGH Alone
Drug: Increlex® (Mecasermin [rDNA origin] injection) + NutropinAq® (Somatropin [rDNA origin]) — rhGH 45µg/kg and rhIGF-1 150µg/kg once daily injection
  Other Names: Increlex; rhIGF-1; GH
  Arms: 4. Combination Dose
Drug: Increlex® (Mecasermin [rDNA origin] injection) + NutropinAq® (Somatropin [rDNA origin]) — rhGH (Somatropin) 45µg/kg and rhIGF-1 (Mecasermin) 50µg/kg once daily injections
  Other Names: Increlex; rhIGF-1; GH
  Arms: 2. Combination Dose
Drug: Increlex® (Mecasermin [rDNA origin] injection) + NutropinAq® (Somatropin [rDNA origin]) — rhGH 45µg/kg and rhIGF-1 100µg/kg once daily injections
  Other Names: Increlex; rhIGF-1; GH
  Arms: 3. Combination Dose

SUMMARY:
IGF-1 (insulin-like growth factor-1) is a hormone that is normally produced in the body in response to another hormone called growth hormone. Growth Hormone is produced by a small gland at the base of the brain (the pituitary). Together IGF-1 and GH are large contributors to growth during infancy, childhood, and adolescence.

Children with IGF Deficiency are short and have an imbalance in the levels of growth hormone and IGF-1 that their body produces. Their growth hormone levels are normal or even high, but IGF-1 levels do not increase normally in response to growth hormone. As a result, they have a type of growth hormone insensitivity and an inability to grow normally.

This study is a test to see whether daily dosing with a combination of rhIGF-1 and rhGH will help children with IGFD grow taller more quickly than children treated with rhGH alone. The study medications, rhIGF-1 and rhGH, are approved by the US Food and Drug Administration (FDA) for use in some growth disorders in children, but the combination of rhIGF-1 and rhGH in children with IGF-1 deficiency (IGFD) is investigational.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legally authorized representatives must give signed informed consent before any trial-related activities
* IGF-1 SDS of ≤ -1 for age and gender
* Short stature, as defined by a height SDS of ≤ -2 for age and gender
* Chronological age ≥ 5 years
* Bone age ≤ 11 years in boys and ≤ 9 years in girls
* GH sufficiency, defined as a maximal stimulated GH response of greater than or equal to 10 ng/mL at Visit 2 (note: upon approval of the Medical Monitor, the result of a prior GH stimulation test may satisfy this requirement).
* Prepubertal status
* Adequate nutrition as evidenced by a body mass index (BMI) greater than or equal to the 5th percentile for age and gender

Exclusion Criteria:

* Severe Primary IGFD (defined as height and IGF-1 SDS ≤ 3, and stimulated GH response greater than or equal to 10 ng/mL)
* Prior or current use of medications with the potential to alter growth patterns including GH, IGF-1, IGFBP-3, gonadotrophin agonists (e.g., Lupron), aromatase inhibitors, androgens and estrogens
* Known or suspected allergy to rhGH, rhIGF-1 or a constituent of their formulations
* Current use of medications for attention deficit disorder
* A chronic health condition that requires anti-inflammatory steroids or daily medication unless approved by the Medical Monitor

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen (formerly Tercica, Inc.)
Locations (1):
- Ipsen, Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrolment: December 2007. Date of last completed: March 2012. This was a Phase II, multicenter, randomized, open-label, parallel-group, active treatment controlled, dose selection study conducted at 27 centers in the US.
Pre-assignment Details: Study screened 155 subjects. Due to failure in screening 49 subjects were excluded from the trial before assignment to groups.
Groups:
- 45 rhGH Alone: Nutropin AQ® (Somatropin [rDNA origin]): Recombinant Human Growth Hormone (rhGH) (Somatropin) 45µg/kg once daily injection
- 45 rhGH + 50 rhIGF-1: Increlex® (Mecasermin [rDNA origin] injection) + Nutropin AQ® (Somatropin [rDNA origin]): rhGH (Somatropin) 45µg/kg and Recombinant Human Insulin-Like Growth Factor-1 (rhIGF-1) (Mecasermin) 50µg/kg once daily injections
- 45 rhGH + 100 rhIGF-1: Increlex® (Mecasermin [rDNA origin] injection) + Nutropin AQ® (Somatropin [rDNA origin]): rhGH 45µg/kg and rhIGF-1 100µg/kg once daily injections
- 45 rhGH + 150 rhIGF-1: Increlex® (Mecasermin [rDNA origin] injection) + Nutropin AQ® (Somatropin [rDNA origin]): rhGH 45µg/kg and rhIGF-1 150µg/kg once daily injection
Period: Overall Study
Arm/Group | 45 rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Started | 26 | 27 | 27 | 26
Completed | 0 | 1 | 0 | 1
Not Completed | 26 | 26 | 27 | 25
Not completed — Adverse Event | 3 | 1 | 5 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 2
Not completed — Patient/Parent Decision | 1 | 6 | 4 | 3
Not completed — Sponsor Decision | 20 | 16 | 17 | 19

BASELINE CHARACTERISTICS:
Population: All Subjects
Groups:
- 45 rhGH Alone: Nutropin AQ® (Somatropin [rDNA origin]): rhGH (Somatropin) 45µg/kg once daily injection
- 45 rhGH + 50 rhIGF-1: Increlex® (Mecasermin [rDNA origin] injection) + Nutropin AQ® (Somatropin [rDNA origin]): rhGH (Somatropin) 45µg/kg and rhIGF-1 (Mecasermin) 50µg/kg once daily injections
- Total: Total of all reporting groups
Arm/Group | 45 rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1 | Total
Number analyzed (Participants) | 26 | 27 | 27 | 26 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (2.0) | 8.4 (2.0) | 9.0 (2.2) | 8.8 (2.3) | 8.8 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 4 | 21
  Male | 21 | 22 | 20 | 22 | 85
Race [Number; unit: participants]
  Asian | 2 | 4 | 1 | 1 | 8
  Black | 1 | 1 | 1 | 0 | 3
  Hispanic | 4 | 1 | 3 | 2 | 10
  White | 17 | 20 | 19 | 23 | 79
  Hispanic/White | 1 | 1 | 3 | 0 | 5
  Hawaiian or Pacific Islander/ White | 1 | 0 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: Standard Deviation Score (SDS)] — Height was measured standing and without shoes, and recorded as the mean of three measurements (the subject being repositioned each time) by the same observer using a Harpenden or other wall-mounted stadiometer which was to be calibrated prior to measurement of each subject and a calibration log kept.
  The SDS calculation and description is specified in baseline characteristic for parameter 'Weight'
  Standard Deviation Score (SDS) | -2.5 (0.5) | -2.5 (0.4) | -2.6 (0.4) | -2.6 (0.4) | -2.5 (0.4)
Weight [Mean (Standard Deviation); unit: SDS] — Weight was recorded from a single observation of the subject in light clothing or dressing gown with shoes removed.
  The SDS was calculated as: SDS=[(value /M)^L - 1] / LS; using power (L), Mean (M) and coefficient of variation (S). The reference values were dependent on gender in addition to age and were selected at the age the closest below subject's age. SDS scores were calculated using L, M and S as defined in the National Center for Health Statistics 2000 data as provided by the Center for Disease Control (Kuczmarski, Ogden et al. 2002)
  SDS | -2.0 (0.7) | -2.1 (0.6) | -2.0 (0.7) | -2.2 (0.9) | -2.1 (0.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: SDS] — BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2).
  The SDS was calculated as: SDS=[(value /M)^L - 1] / LS; using power (L), Mean (M) and coefficient of variation (S). The reference values were dependent on gender in addition to age and were selected at the age the closest below subject's age. SDS scores were calculated using L, M and S as defined in the National Center for Health Statistics 2000 data as provided by the Center for Disease Control (Kuczmarski, Ogden et al. 2002)
  SDS | -0.3 (0.7) | -0.5 (0.7) | -0.4 (0.7) | -0.5 (0.8) | -0.4 (0.7)
IGF-1 [Mean (Standard Deviation); unit: SDS] — IGF-1 SDS was computed based on actual value of IGF-1, the mean reference value of IGF-1 and the SD reference value of IGF-1 as defined in the International Congress of Endocrinology, Lisbon, 2004
  SDS | -1.8 (0.5) | -2.0 (0.7) | -1.8 (0.6) | -2.0 (0.6) | -1.9 (0.6)
Mid-Parental target height [Mean (Standard Deviation); unit: SDS] — The mid-parental target height SDS is defined as: 0.4*(Mother's Height SDS+Father's Height SDS)
  The SDS was calculated as: SDS=[(value /M)^L - 1] / LS; using power (L), Mean (M) and coefficient of variation (S). The reference values were dependent on gender in addition to age and were selected at the age the closest below subject's age. SDS scores were calculated using L, M and S as defined in the National Center for Health Statistics 2000 data as provided by the Center for Disease Control (Kuczmarski, Ogden et al. 2002)
  SDS | -0.5 (0.4) | -0.6 (0.5) | -0.5 (0.5) | -0.5 (0.5) | -0.5 (0.5)
Bone age imputed [Mean (Standard Deviation); unit: years] | 7.6 (1.7) | 7.2 (1.8) | 7.2 (2.0) | 7.3 (2.0) | 7.3 (1.9)
Height Age [Mean (Standard Deviation); unit: years] | 6.5 (1.6) | 6.0 (1.5) | 6.4 (1.8) | 6.2 (1.9) | 6.3 (1.7)
Max stimulated GH [Mean (Standard Deviation); unit: ng/mL] | 17.9 (8.9) | 18.2 (8.4) | 19.5 (6.3) | 20.1 (8.4) | 18.9 (8.0)
IGFBP-3 SDS [Mean (Standard Deviation); unit: SDS] — Number of subjects analysed= 26,26,27,26 (Total 105)
  IGFBP-3 SDS was computed based on actual value of IGFBP-3, the mean reference value of IGFBP-3 and the SD reference value of IGFBP-3 as defined in the International Congress of Endocrinology, Lisbon, 2004
  SDS | -1.1 (0.7) | -1.2 (0.9) | -1.0 (0.8) | -1.3 (0.8) | -1.1 (0.8)
Mother height [Mean (Standard Deviation); unit: cm] — Number of subjects analysed= 24,23,25,25 (Total 97)
  cm | 157 (5) | 157 (5) | 157 (6) | 159 (7) | 158 (6)
Father height [Mean (Standard Deviation); unit: cm] — Number of subjects analysed= 18,20,22,21 (Total = 81)
  cm | 172 (4) | 169 (5) | 173 (7) | 172 (6) | 172 (6)

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity
Time Frame: First year of treatment
Population: Modified Intent-To-Treat (MITT): MITT population comprised all subjects who were randomized and had at least one post-baseline height measurement.
  [n= 25,27,27,26]
Measure: Mean (Standard Deviation); unit: cm/y
Groups:
- rhGH Alone: Nutropin AQ® (Somatropin [rDNA origin]): rhGH (Somatropin) 45µg/kg once daily injection
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
cm/y | 9.3 (1.7) | 10.1 (1.3) | 9.7 (2.5) | 11.2 (2.1)

2. Secondary Outcome: Height Velocity
Time Frame: Second, third and fourth year
Population: Modified Intent-To-Treat (MITT): MITT population comprised all subjects who were randomized and had at least one post-baseline height measurement.
Measure: Mean (Standard Deviation); unit: cm/y
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
cm/y
  Year 2 height velocity [n= 24,25,22,24] | 8.4 (1.3) | 9.1 (1.2) | 9.4 (1.6) | 10.1 (1.8)
  Year 3 height velocity [n= 22,22,20,22] | 8.0 (1.1) | 8.4 (1.0) | 8.9 (1.3) | 9.2 (1.5)
  Year 4 height velocity [n= 17,16,15,16] | 7.7 (0.9) | 8.1 (0.8) | 8.4 (1.2) | 8.3 (1.3)

3. Secondary Outcome: Cumulative Change in Height Standard Deviation Score (SDS)
Description: Height was measured standing and without shoes, and recorded as the mean of three measurements (the subject being repositioned each time) by the same observer using a Harpenden or other wall-mounted stadiometer which was to be calibrated prior to measurement of each subject and a calibration log kept.
  The SDS was calculated as: SDS=[(value /M)^L - 1] / LS; using power (L), Mean (M) and coefficient of variation (S). The reference values were dependent on gender in addition to age and were selected at the age the closest below subject's age. SDS scores were calculated using L, M and S as defined in the National Center for Health Statistics 2000 data as provided by the Center for Disease Control (Kuczmarski, Ogden et al. 2002)
Time Frame: First, second, third and fourth year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
SDS
  First year [n= 25,27,27,26] | 0.7 (0.3) | 0.9 (0.2) | 0.8 (0.4) | 1.0 (0.4)
  Second year [n= 24,25,22,24] | 1.0 (0.4) | 1.4 (0.4) | 1.4 (0.5) | 1.6 (0.6)
  Third year [n=22,22,20,22] | 1.3 (0.5) | 1.6 (0.4) | 1.8 (0.7) | 1.9 (0.6)
  Fourth year [n=17,16,15,16] | 1.5 (0.5) | 1.8 (0.5) | 2.1 (0.8) | 2.0 (0.7)

4. Secondary Outcome: Predicted Adult Height (PAH)
Description: Predicted Adult Height calculated by method, Roche-Wainer-Thissen (RWT) and mid-parental target height SDS.
  The SDS was calculated as: SDS=[(value /M)^L - 1] / LS; using power (L), Mean (M) and coefficient of variation (S). The reference values were dependent on gender in addition to age and were selected at the age the closest below subject's age. SDS scores were calculated using L, M and S as defined in the National Center for Health Statistics 2000 data as provided by the Center for Disease Control (Kuczmarski, Ogden et al. 2002)
Time Frame: At baseline (Day 1), year 1,2,3 and 4
Population: Completers, the completer population consists of all subjects that remained in the study until a specific time point (ie; Year 1, Year 2, Year 3 and Year 4).
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
SDS
  Baseline (day 1) [n=25,27,27,26] | -1.67 (0.51) | -1.83 (0.58) | -1.69 (0.59) | -1.76 (0.73)
  Year 1 [n= 24,25,22,25] | -1.12 (0.57) | -1.22 (0.58) | -0.99 (0.55) | -1.01 (0.80)
  Year 2 [n= 22,21,20,22] | -0.96 (0.56) | -0.81 (0.55) | -0.66 (0.56) | -0.69 (0.91)
  Year 3 [n=21,19,19,20] | -0.78 (0.63) | -0.65 (0.60) | -0.42 (0.62) | -0.64 (0.98)
  Year 4 [n=3,4,4,3] | -1.22 (0.59) | -0.44 (0.81) | 0.49 (0.60) | -0.07 (0.89)
  Mid-parental target height [n=25,27,27,26] | -0.51 (0.38) | -0.64 (0.52) | -0.53 (0.50) | -0.47 (0.51)

5. Secondary Outcome: Total Change From Baseline (Day 1) in BMI SDS
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2).
  The SDS was calculated as: SDS=[(value /M)^L - 1] / LS; using power (L), Mean (M) and coefficient of variation (S). The reference values were dependent on gender in addition to age and were selected at the age the closest below subject's age. SDS scores were calculated using L, M and S as defined in the National Center for Health Statistics 2000 data as provided by the Center for Disease Control (Kuczmarski, Ogden et al. 2002)
Time Frame: At year 1,2,3,4 and end of study (visit 23) versus baseline (day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
SDS
  Change from day 1 to year 1 [n= 24,25,22,25] | 0.24 (0.43) | 0.31 (0.39) | 0.36 (0.41) | 0.54 (0.40)
  Change from day 1 to year 2 [n= 22,21,20,22] | 0.31 (0.49) | 0.57 (0.41) | 0.49 (0.44) | 0.59 (0.46)
  Change from day 1 to year 3 [n=21,19,19,20] | 0.35 (0.58) | 0.62 (0.43) | 0.49 (0.59) | 0.71 (0.54)
  Change from day 1 to year 4 [n=3,5,5,4] | 0.27 (0.52) | 0.64 (0.58) | 0.65 (0.90) | 1.20 (0.91)
  Change from day 1 to visit 23 [n=25,27,27,26] | 0.34 (0.54) | 0.45 (0.45) | 0.42 (0.53) | 0.64 (0.60)

6. Secondary Outcome: Skeletal Maturation
Description: Assessed by bone age. Bone age was determined by the radiograph.
  The SDS was calculated as: SDS=[(value /M)^L - 1] / LS; using power (L), Mean (M) and coefficient of variation (S). The reference values were dependent on gender in addition to age and were selected at the age the closest below subject's age. SDS scores were calculated using L, M and S as defined in the National Center for Health Statistics 2000 data as provided by the Center for Disease Control (Kuczmarski, Ogden et al. 2002)
Time Frame: At baseline(day 1), year 1,2,3 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
SDS
  Baseline [n=25,27,27,26] | 7.6 (1.8) | 7.3 (1.9) | 7.2 (2.0) | 7.4 (2.0)
  Year 1 [n= 24,25,22,25] | 9.0 (1.9) | 8.5 (1.9) | 8.4 (2.2) | 8.5 (2.1)
  Year 2 [n= 22,21,20,22] | 10.3 (2.0) | 9.6 (2.1) | 9.8 (2.4) | 9.9 (2.2)
  Year 3 [n=21,19,19,20] | 11.4 (2.0) | 10.9 (2.2) | 11.4 (2.4) | 10.9 (2.2)
  Year 4 [n=3,4,5,3] | 12.4 (1.0) | 10.9 (1.8) | 12.2 (3.0) | 12.5 (2.1)

7. Secondary Outcome: Changes From Baseline (Day 1) in Serum Concentrations of Growth Hormone (GH)
Time Frame: At Baseline (Day 1), Year 1,2,3 and 4
Population: Modified Intent-to-Treat (MITT) Population comprised all subjects who were randomized and had at least one post-baseline height measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
ng/mL
  Day 1 (Baseline) [n=23,25,18,25] | 1.1 (2.2) | 2.9 (8.1) | 2.4 (4.5) | 1.9 (2.3)
  Year 1 (Trough) [n=23,25,18,25] | 1.7 (2.1) | 3.5 (12.9) | 2.1 (3.2) | 1.4 (2.1)
  Year 2 (Trough) [n=21,20,16,20] | 4.0 (6.0) | 2.2 (4.2) | 2.7 (3.9) | 1.4 (1.2)
  Year 3 (Trough) [n=20,18,15,20] | 2.8 (5.1) | 1.3 (1.6) | 1.5 (1.4) | 1.9 (3.5)
  Year 4 (Trough) [n=3,5,4,3] | 1.2 (0.3) | 0.5 (0.4) | 3.0 (2.9) | 1.1 (0.6)

8. Secondary Outcome: Changes From Baseline (Day 1) in Serum Concentrations of Insulin-Like Growth Factor-1 (IGF-1)
Time Frame: At Baseline (Day 1), Year 1,2,3 and 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
ng/mL
  Day 1 (Baseline) [n= 24,25,22,25] | 108.3 (39.8) | 87.1 (31.0) | 100.2 (41.4) | 96.7 (38.8)
  Year 1 (Trough) [n= 24,25,22,25] | 278.2 (95.5) | 326.9 (108.9) | 397.8 (185.4) | 296.0 (126.8)
  Year 2 (Trough) [n= 22,21,20,22] | 312.8 (97.2) | 427.2 (178.5) | 539.3 (195.9) | 466.4 (178.6)
  Year 3 (Trough)[n= 21,19,19, 20] | 335.3 (110.0) | 404.9 (104.4) | 462.2 (156.4) | 441.3 (226.0)
  Year 4 (Trough)[n= 3,5,5,3] | 347.7 (130.7) | 363.6 (125.4) | 546.2 (265.8) | 607.7 (65.0)

9. Secondary Outcome: Changes From Baseline (Day 1) in Serum Concentrations of Insulin-Like Growth Factor Binding Protein-1 (IGFBP-1)
Time Frame: At Baseline (Day 1), Year 1,2,3 and 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
ng/mL
  Day 1 (Baseline) [n= 24,24,21,24] | 87.8 (54.5) | 102.5 (37.2) | 95.7 (50.0) | 122.4 (53.7)
  Year 1 (Trough) [n= 24,24,21,24] | 45.7 (38.0) | 63.8 (50.1) | 68.2 (61.6) | 88.8 (47.4)
  Year 2 (Trough) [n= 22,21,19,20] | 59.4 (45.6) | 58.2 (47.7) | 53.3 (35.3) | 71.7 (46.1)
  Year 3 (Trough) [n= 21,19,18,19] | 46.1 (35.2) | 60.4 (52.5) | 53.2 (34.8) | 84.7 (53.5)
  Year 4 (Trough) [n= 3,5,5,3] | 100.0 (60.4) | 46.8 (58.0) | 49.2 (20.7) | 49.0 (26.9)

10. Secondary Outcome: Changes From Baseline (Day 1) in Serum Concentrations of Insulin-Like Growth Factor Binding Protein-3 (IGFPB-3)
Time Frame: At Baseline (Day 1), Year 1,2,3 and 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
ng/mL
  Day 1 (Baseline) [n= 24,25,22,25] | 2204.2 (387.3) | 2160.0 (421.3) | 2113.6 (486.3) | 2196.0 (612.0)
  Year 1 (Trough) [n= 24,25,22,25] | 2954.2 (618.5) | 2784.0 (755.9) | 2677.3 (548.5) | 2624.0 (598.8)
  Year 2 (Trough) [n= 22,21,20,22] | 2813.6 (399.2) | 2942.9 (552.8) | 3060.0 (703.7) | 2754.5 (600.6)
  Year 3 (Trough) [n= 21,19,19,20] | 3404.8 (476.9) | 3431.6 (718.1) | 3373.7 (479.4) | 3260.0 (908.1)
  Year 4 (Trough) [n= 3,5,5,3] | 3733.3 (378.6) | 3260.0 (709.2) | 3620.0 (957.6) | 3466.7 (461.9)

11. Secondary Outcome: Changes From Baseline (Day 1) in Serum Concentrations of Acid-Labile Subunit (ALS)
Time Frame: At Baseline (Day 1), Year 1,2,3 and 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
mg/L
  Day 1 (Baseline) [n=25,26,26,25] | 10.6 (3.0) | 10.0 (3.4) | 10.9 (3.0) | 11.0 (4.1)
  Year 1 (Trough) [n=24,24,21,24] | 16.0 (4.0) | 12.7 (2.3) | 14.0 (3.9) | 11.5 (2.8)
  Year 2 (Trough) [n= 22,21,19,20] | 15.2 (4.3) | 14.3 (5.2) | 15.7 (4.0) | 13.7 (4.5)
  Year 3 (Trough) [n= 21,18,18,19] | 13.7 (2.3) | 13.0 (3.2) | 12.9 (2.7) | 11.2 (4.0)
  Year 4 (Trough) [n= 3,5,5,3] | 13.7 (1.5) | 12.0 (2.2) | 12.0 (3.0) | 13.7 (2.1)

12. Secondary Outcome: Changes From Baseline (Day 1) in Serum Concentrations of Growth Hormone Binding Protein (GHBP)
Time Frame: At Baseline (Day 1), Year 1,2,3 and 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 25 | 27 | 27 | 26
pmol/L
  Day 1 (Baseline) [n= 25,26,25,25] | 785.8 (291.1) | 735.8 (343.5) | 698.8 (212.2) | 719.0 (261.5)
  Year 1 (Trough) [n= 23,24,20,24] | 729.4 (229.5) | 576.9 (211.0) | 598.9 (187.3) | 530.5 (233.5)
  Year 2 (Trough) [n=22,21,18,21] | 725.6 (308.4) | 589.3 (171.6) | 562.5 (184.4) | 564.6 (171.9)
  Year 3 (Trough) [n= 21,17,17,19] | 672.0 (224.4) | 646.9 (204.1) | 614.3 (210.9) | 554.9 (197.0)
  Year 4 (Trough) [n= 3,5,5,3] | 714.0 (38.5) | 516.9 (252.5) | 798.2 (336.1) | 519.7 (141.1)

13. Secondary Outcome: Summary of Adverse Events With Number of Occurrences
Description: A Data Monitoring Committee (DMC) was established to monitor subject safety
Time Frame: Approximately up to 4 years.
Population: Safety population: Safety population consisted of all subjects who were randomized. Note that post baseline follow-up data were received for all subjects who were randomized.
Measure: Number; unit: Number of events
Arm/Group | rhGH Alone | 45 rhGH + 50 rhIGF-1 | 45 rhGH + 100 rhIGF-1 | 45 rhGH + 150 rhIGF-1
Number analyzed (Participants) | 26 | 27 | 27 | 26
Number of events
  Any Adverse Event | 381 | 416 | 401 | 518
  Any TEAE | 374 | 406 | 392 | 513
  Severe TEAEs | 5 | 5 | 3 | 3
  Moderate TEAE | 60 | 55 | 57 | 86
  Mild TEAE | 309 | 346 | 332 | 424
  Related TEAEs | 27 | 53 | 74 | 119
  Related and Severe | 1 | 1 | 1 | 0
  Related and Moderate | 5 | 4 | 18 | 13
  Related and Mild | 21 | 48 | 55 | 106
  TEAEs Leading to Study Withdrawal | 18 | 17 | 36 | 6
  SAEs | 1 | 6 | 2 | 1
  Deaths | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximate up to 4 years
Description: Treatment emergent adverse event (TEAEs) Reported in ≥5% Subjects Receiving rhGH Alone or Receiving Combination Therapy.
  Safety population consisted of all subjects who were randomized. Note that post baseline follow-up data were received for all subjects who were randomized.
Groups:
- 1. rhGH Alone: Nutropin AQ® (Somatropin [rDNA origin]): rhGH (Somatropin) 45µg/kg once daily injection
- 2. 45 rhGH + 50 rhIGF-1: Increlex® (Mecasermin [rDNA origin] injection) + Nutropin AQ® (Somatropin [rDNA origin]): rhGH (Somatropin) 45µg/kg and rhIGF-1 (Mecasermin) 50µg/kg once daily injections
- 3. 45 rhGH + 100 rhIGF-1: Increlex® (Mecasermin [rDNA origin] injection) + Nutropin AQ® (Somatropin [rDNA origin]): rhGH 45µg/kg and rhIGF-1 100µg/kg once daily injections
- 4. 45 rhGH + 150 rhIGF-1: Increlex® (Mecasermin [rDNA origin] injection) + Nutropin AQ® (Somatropin [rDNA origin]): rhGH 45µg/kg and rhIGF-1 150µg/kg once daily injection
Arm/Group | 1. rhGH Alone | 2. 45 rhGH + 50 rhIGF-1 | 3. 45 rhGH + 100 rhIGF-1 | 4. 45 rhGH + 150 rhIGF-1
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/27 | 2/27 | 1/26
Other Adverse Events (participants affected / at risk) | 26/26 | 27/27 | 27/27 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. rhGH Alone (N=26) | 2. 45 rhGH + 50 rhIGF-1 (N=27) | 3. 45 rhGH + 100 rhIGF-1 (N=27) | 4. 45 rhGH + 150 rhIGF-1 (N=26)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Evans syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. rhGH Alone (N=26) | 2. 45 rhGH + 50 rhIGF-1 (N=27) | 3. 45 rhGH + 100 rhIGF-1 (N=27) | 4. 45 rhGH + 150 rhIGF-1 (N=26)
Upper respiratory tract infection (Infections and infestations) | 10 (23) | 10 (19) | 9 (31) | 13 (37)
Otitis media (Infections and infestations) | 4 (4) | 5 (7) | 3 (5) | 9 (19)
Viral infection (Infections and infestations) | 6 (10) | 3 (7) | 6 (6) | 8 (21)
Gastroenteritis (Infections and infestations) | 1 (2) | 3 (3) | 5 (9) | 6 (10)
Pharyngitis streptococcal (Infections and infestations) | 5 (13) | 12 (17) | 7 (9) | 6 (14)
Gastroenteritis viral (Infections and infestations) | 6 (8) | 3 (9) | 2 (4) | 4 (4)
Influenza (Infections and infestations) | 2 (2) | 3 (4) | 5 (6) | 4 (4)
Ear infection (Infections and infestations) | 3 (5) | 2 (4) | 4 (6) | 3 (4)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Molluscum contagiosum (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (3) | 2 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 4 (5) | 4 (15) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 5 (25) | 7 (14) | 3 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (17) | 5 (6) | 6 (12) | 12 (19)
Abdominal pain upper (Infections and infestations) | 7 (11) | 5 (8) | 3 (7) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (10) | 4 (5) | 4 (7) | 6 (11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (6) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (4)
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 9 (17) | 15 (27) | 4 (22) | 13 (19)
Injection site pain (General disorders) | 4 (4) | 1 (2) | 0 (0) | 4 (6)
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Injection site bruising (General disorders) | 4 (4) | 4 (5) | 4 (4) | 3 (5)
Injection site hypertrophy (General disorders) | 0 (0) | 6 (8) | 7 (13) | 3 (4)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Injection site urticaria (General disorders) | 2 (3) | 3 (3) | 1 (2) | 2 (5)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 14 (40) | 14 (43) | 17 (39) | 18 (50)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4) | 0 (0) | 2 (3)
Migraine (Nervous system disorders) | 1 (2) | 3 (3) | 3 (3) | 1 (7)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (6)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (6) | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 1 (2) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Orthodontic appliance complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 14 (18) | 9 (16) | 10 (14)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (11) | 7 (10) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (6) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 1 (1) | 1 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (7) | 5 (5) | 6 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 8 (11) | 7 (8) | 5 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5) | 1 (1) | 4 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2) | 3 (4) | 3 (3) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Insulin-like growth factor increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Body temperature increased (Investigations) | 1 (1) | 3 (4) | 3 (3) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (3) | 4 (5)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Attention (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (7) | 1 (1) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Enuresis (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated once the last subject had completed three years of treatment (compared to the six years planned in protocol Amendment) for strategic reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less